CLINICAL TRIAL: NCT06435013
Title: Lenvatinib Versus Bevacizumab Combined With Immune Checkpoint Inhibitors and Hepatic Arterial Infusion Chemotherapy in Unresectable Hepatocellular Carcinoma: A Retrospective, Multi-center, and Propensity Score Matching Study
Brief Title: Lenvatinib vs Bevacizumab Plus ICIs and HAIC in Unresectable HCC
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Ming Shi, Sun Yat-sen University
Other Study IDs: LenBev-001
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LenHAP: Lenvatinib combined with hepatic arterial infusion chemotherapy and PD-1/PD-L1;
  Interventions: Drug: Lenvatinib
- BevHAP: Bevacizumab combined with hepatic arterial infusion chemotherapy and PD-1/PD-L1;

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib combined with hepatic arterial infusion chemotherapy and PD-1/PD-L1;
  Groups: LenHAP

SUMMARY:
Previous studies had suggested hepatic arterial infusion chemotherapy (HAIC) combined with immune checkpoint inhibitors (ICIs) and anti-angiogenic drugs had promising anti-tumor activity in unresectable hepatocellular carcinoma (HCC). Two kinds of anti-angiogenic drugs (tyrosine kinase inhibitors [lenvatinib] and anti-VEGF antibody [bevacizumab]) were applied in first-line treatment of unresectable HCC. However, little is known about the difference of efficacy and safety between lenvatinib (LenHAP) or bevacizumab (BevHAP) combined with ICIs and HAIC in unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:patients aged 18 years or older, with unresectable, locally advanced, or metastatic HCC, with the diagnosis confirmed by histologic or cytologic analysis or clinical features according to the American Association for the Study of Liver Disease criteria(15), who had received no previous treatment, had at least on measurable disease, as defined by Response Evaluation Criteria In Solid Tumours version 1.1 (RECIST v1.1) criteria(16), had a baseline Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, had a Child-Pugh liver function score of 7 or less and had adequate hematologic and organ function (absolute neutrophil count ≥1.2×109/l, platelet count ≥60×109/l, total bilirubin <30μmol/l, albumin ≥30g/l, aspartate transaminase and alanine transaminase ≤5×upper limit of the normal, creatinine clearance rate of ≤1.5×upper limit of the normal, and left ventricular ejection ≥45%) -

Exclusion Criteria:history of HIV, organ allograft, combined with other malignant tumors, evidence of hepatic decompensation, bleeding diathesis or event, and allergy to the investigational agents or any agent given in association with this trial and incomplete medical information.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with received the combination therapy of lenvatinib/bevacizumab, hepatic arterial infusion chemotherapy and PD-1/L1
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
progression-free survival | 2015-1 to 2023-4

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No